CLINICAL TRIAL: NCT00004845
Title: A Multicenter Trial of Rofecoxib and Naproxen in Alzheimer's Disease
Brief Title: A Multicenter Trial of Rofecoxib and Naproxen in Alzheimer's Disease (NSAID Study)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: IA0021
Record Dates: First submitted 2000-02-28; First posted 2000-02-29 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-06

CONDITIONS: Alzheimer Disease
Keywords: Anti-inflammatory
MeSH Terms: conditions — Alzheimer Disease | interventions — rofecoxib; Naproxen

INTERVENTIONS:
Drug: Rofecoxib
Drug: Naproxen

SUMMARY:
The primary specific aim of this clinical trial is to determine whether treatment with rofecoxib or naproxen for one year will slow the rate of decline of cognitive function in patients with Alzheimer's disease (AD) as measured by ADAScog.

DETAILED DESCRIPTION:
Evidence that inflammatory mechanisms contribute to neuronal injury in Alzheimer's disease along with a number of epidemiological studies suggests that non-steroidal anti-inflammatory drugs (NSAIDs) may slow the rate of cognitive deterioration. We have selected two such drugs for a therapeutic trial: rofecoxib and naproxen. The trial employs a double-blind parallel design with three primary treatment groups: rofecoxib, naproxen and placebo. A total of 320 patients will be enrolled in the trial and randomized to the three groups. Stable use of cholinesterase inhibitors, estrogen, low dose aspirin, and vitamin E will be allowed. Patients with inflammatory diseases that might respond to the study medications will be excluded.

The primary outcome measure will be the one year change in the cognitive subscale of the Alzheimer's Disease Assessment Scale (ADAScog). The attainment of significant endpoints will be examined as a secondary outcome measure. Other secondary measures include the CDR sum-of-boxes, Neuropsychiatric Inventory, the Quality of Life-AD and the ADCS pharmacoeconomic scale. The influence of HLA-DR (Human Leukocyte Antigen) genotype on clinical progression and response to treatment will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* NINCDS/ADRDA criteria for probable AD
* MMSE between 13 and 26, inclusive
* Stable medical condition for 3 months
* Screening visit
* Physically acceptable for this study as confirmed by medical history, physical exam, neurologic exam, and clinical laboratory tests
* Supervision available for administration of study medications; caregiver/informant to accompany patient to all scheduled visits
* Fluent in English or Spanish
* Age greater than or equal to 55 years old
* Modified Hachinski of less than or equal to 4
* CT or MRI since onset of memory impairment demonstrating absence of clinically significant focal lesion
* Able to complete baseline assessments
* 6 years of education or work history sufficient to exclude mental retardation
* Able to ingest oral medication

Exclusion Criteria:

* Hypersensitivity to aspirin or NSAID
* Active peptic ulcer disease within 5 years
* Renal insufficiency with creatinine greater than 1.5
* Clinically significant liver disease
* Poorly controlled hypertension
* Congestive heart failure
* Bleeding ulcer
* Active neoplastic disease (skin tumors other than melanoma are not exclusionary; patients with stable prostate cancer may be included at the discretion of the project director)
* Inflammatory diseases (including crystal arthropathy, rheumatoid arthritis, systemic lupus, erythematosus, Sjogren's syndrome, inflammatory bowel disease)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon Thal, MD, Principal Investigator — Alzheimer's Disease Cooperative Study
Locations (40):
- United States (40):
  - Barrow Neurological Group, Phoenix, Arizona
  - University of Arizona, Tucson, Tucson, Arizona
  - University of California Irvine Institute for Brain Aging and Dementia, Irvine, California
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Davis, Martinez, California
  - Yale University, School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Baumel-Eisner Neuromedical Institute, Boca Raton, Boca Raton, Florida
  - Baumel-Eisner Ft Lauderdale, Fort Lauderdale, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Wein Center, Miami Beach, Florida
  - Baumel-Eisner Neuromedical Institute, MiamiBeach, Miami Beach, Florida
  - University of South Florida, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Rush Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Kansas University, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nevada, Las Vegas, Nevada
  - ClinSearch, Inc, Summit, New Jersey
  - New York University Medical Center, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Memorial Hospital of Rhode Island, Providence, Rhode Island
  - Medical University of South Carolina, North Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas, SW Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Aisen PS, Schafer KA, Grundman M, Pfeiffer E, Sano M, Davis KL, Farlow MR, Jin S, Thomas RG, Thal LJ; Alzheimer's Disease Cooperative Study. Effects of rofecoxib or naproxen vs placebo on Alzheimer disease progression: a randomized controlled trial. JAMA. 2003 Jun 4;289(21):2819-26. doi: 10.1001/jama.289.21.2819. PMID 12783912